CLINICAL TRIAL: NCT03636997
Title: Treatment of Complex Anal Fistula With Draining Seton With or Without Rerouting of the Fistula Track: a Randomized Controlled Trial
Brief Title: Treatment of Complex Anal Fistula With Draining Seton With or Without Rerouting of Track
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of general surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mansoura63
Record Dates: First submitted 2018-08-16; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Draining seton (Active Comparator): Draining seton is placed through the fistula track and internal and external anal sphicnters
  Interventions: Procedure: Draining seton
- Rerouting of track (Active Comparator): The seton and the fistula track are rerouted to include the internal anal sphincter only and spare the external anal sphincter
  Interventions: Procedure: Rerouting of track

INTERVENTIONS:
Procedure: Draining seton — Number 1 silk suture was passed through the fistula track and tied as loose seton
  Arms: Draining seton
Procedure: Rerouting of track — The seton and fistula track were rerouted to involve the internal anal sphicnter only and spare the external sphincter
  Arms: Rerouting of track

SUMMARY:
This randomized trial aimed to compare conventional draining seton with or without rerouting of the fistula track in treatment of complex anal fistula

DETAILED DESCRIPTION:
Placement of seton is typically employed when the fistula track is involving more than 30% of the external anal sphincter. However, attempts to reroute the seton and the involved fistula track were made to preserve the external anal sphincter fibers and hasten healing of the anal wound. Mann and Clifton first introduced a transposition technique for the management of high anal and anorectal fistulas by re-routing the extrasphincteric portion of the track into an intersphincteric position with immediate repair of the external sphincter and reported successful outcomes of five patients in terms of quick healing and preserved anal continence.

The present study aimed to evaluate the outcome of draining seton with or without rerouting of the fistula track in treatment complex high anal fistula regarding healing time, postoperative pain, and incidence of recurrence and FI postoperatively. We hypothesized that rerouting the seton to include the fistula track and the internal anal sphincter only, preserving the external anal sphincter muscles, would serve to hasten healing and decrease the incidence of recurrence and continence disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both genders aging below 60 years old with complex crypto-glandular anal fistula were included. Complex anal fistula were defined as high trans-sphincteric anal fistulas involving more than 30% of the external anal sphincter fibers, suprasphincteric, extrasphincteric, and horse-shoe fistula

Exclusion Criteria:

* Patients with simple anal fistula.
* Patients with acute anorectal sepsis.
* Patients with secondary anal fistula caused by inflammatory bowel diseases, sexually transmitted diseases, malignancy, or irradiation.
* Patients with associated anorectal conditions as hemorrhoids, anal fissure, rectal prolapse, or malignancy.
* Patients with history of previous surgical treatment of anal fistula.
* Patients with symptomatic preoperative fecal incontinence.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Healing time | 6 months after surgery
  Time required to achieve complete healing of the anal fistula

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Emile, M.D., Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Omar W, Alqasaby A, Abdelnaby M, Youssef M, Shalaby M, Anwar Abdel-Razik M, Emile SH. Drainage Seton Versus External Anal Sphincter-Sparing Seton After Rerouting of the Fistula Tract in the Treatment of Complex Anal Fistula: A Randomized Controlled Trial. Dis Colon Rectum. 2019 Aug;62(8):980-987. doi: 10.1097/DCR.0000000000001416. PMID 31162376